CLINICAL TRIAL: NCT05924620
Title: Efficacy and Safety of Finerenone in Patients With Primary Aldosteronism: a Randomized, Controlled Trial
Brief Title: Efficacy and Safety of Finerenone in Patients With Primary Aldosteronism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Professor.Qifu Li, Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Finerenone study
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-07

CONDITIONS: Primary Aldosteronism
Keywords: finerenone; spironolactone
MeSH Terms: conditions — Hyperaldosteronism | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Patients with PA using finerenone (Experimental): Patients with PA divided into this group need to take finerenone for 60 days (20mg qd)
  Interventions: Drug: finerenone
- Patients with PA using spironolactone (No Intervention): Patients with PA divided into this group need to take spironolactone for 60 days (20mg qd)

INTERVENTIONS:
Drug: finerenone — Patients with PA divided into Intervention group need to take finerenone for 60 days (20mg qd).
  Other Names: Kerendia
  Arms: Patients with PA using finerenone

SUMMARY:
To study the efficacy and safety of finerenone in patients with primary aldosteronism

DETAILED DESCRIPTION:
This is a prospective and randomized study involving patients with primary aldosteronism(PA). All paticipants will be randomized into finerenone group(Intervention group) and spironolactone group(Control group) and to compare the antihypertensive effect in patients with PA.

If the self-measured blood pressure of patients at home continues to be greater than 140/90 mmHg at 2-4 weeks, spironolactone or finerenone should be increased to 40mg qd, and electrolytes should be reviewed at 2 weeks after dosed.

ELIGIBILITY:
Inclusion Criteria: Patients who meet the following criterion can be included in this study.

1. Patients know the whole process of the trial and voluntarily accepted randomization, intervention and follow-up.
2. Patients voluntarily participated in the study and signed an informed consent, willing to complete all follow-up visits as required.
3. Aged between 18-70, male or female, with legal capacity.
4. eGFR≥60(ml/min/1.73 m2)
5. Patients with PA and substandard blood pressure (≥140/90mmHg) who didn't take any antihypertensive drugs or who had been using antihypertensive drugs other than MRA steadily for 2 weeks or more

Exclusion Criteria: Patients with one of the following conditions will be excluded in this study:

1. To assess patients with poor compliance who had difficulty fully participating in the study, or who refused to sign written informed consent for the study
2. Patients with heart failure (New York Heart Association (NYHA) class III or IV), liver transaminase levels were more than 2 times higher than the upper limit of normal, estimated glomerulus filtration rate<30ml/min/m2
3. Patients with serum potassium > 5.0mmol/L without potassium supplementation
4. Patients with stroke or acute coronary syndrome within 3 months
5. Pregnant or lactating women
6. Patients currently receiving sex hormone or glucocorticoid therapy
7. Patients with a history of uncontrolled malignant tumor
8. Patients who took MRA within 2 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
Compare the change of daytime mean systolic blood pressure in the overall cohort between two groups. | At baseline and 2 month of follow-up
  Measured by ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Compare the serum potassium elevation in the overall cohort between two groups. | At baseline and 2 month of follow-up
  Measured by blood electrolytes
Compare the change of daytime mean diastolic blood pressure in the overall cohort between two groups. | At baseline and 2 month of follow-up
  Measured by ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Q Li, PhD, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No